CLINICAL TRIAL: NCT01557972
Title: Usefulness of Home Blood Pressure Measurement in the Morning in Type 2 Diabetic Patients : Long-term (10 Years) Results of a Prospective Longitudinal Study
Brief Title: Long-term of 10 Years Results of a Prospective Longitudinal Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Nagaoka Red Cross Hospital (Other)
Responsible Party: Principal Investigator, Kyuzi Kamoi, Investigator, Nagaoka Red Cross Hospital
Other Study IDs: 5
Record Dates: First submitted 2012-03-08; First posted 2012-03-20 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Type 2 Diabetes Mellitus; Blood Pressure
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1. Morning HP and NT: Subjects based on HBP were divided into MH and MN patients
  Interventions: Procedure: Blood pressure measurement based on HBP or CBP
- 2. Clinic HP and NT: Subjects based on CBP were divided into CH and CN patients
  Interventions: Procedure: Blood pressure measurement based on HBP or CBP

INTERVENTIONS:
Procedure: Blood pressure measurement based on HBP or CBP — To clarify which of HBP or CBP provides the stronger prediction power for the outcomes.
  Groups: 1. Morning HP and NT
Procedure: Blood pressure measurement based on HBP or CBP — To clarify which of HBP or CBP provides the stronger predictive power for the outcomes
  Groups: 2. Clinic HP and NT

SUMMARY:
Previous cross-sectional studies have demonstrated that blood pressure (BP) measurements at home (HBP) in the morning offer stronger predictive power for micro- and macrovascular complications in patients with type 1 and 2 diabetes than casual/clinic blood pressure measurements (CBP) (Kamoi K et al, 2002-2003). Further, a prospective, longitudinal study for 6 years in patients with type 2 diabetes also demonstrated that control of wakening-up HBP provides the stronger predictive power for the outcomes than that of CBP did (Kamoi et al, 2010).

However, it is not clear to show which of BP measurement provides the stronger predictive power for outcomes by comparing cumulative events over a longer time than 6 years. Therefore, the investigators examined which of HBP or CBP provides the stronger predictive power for outcomes in addition of renal anemia reported previously over 10 years in the patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* After a detailed baseline examination, 400 Japanese subjects with type 2 diabetes reported previously are followed up for all-cause mortality and morbidity.

Exclusion Criteria:

* Other than the above, patients judged inappropriate as the subjects of this study by the investigator

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 400 patients
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 1999-11; Primary Completion 2013-02 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Death | Average time is 10 years
  Number of participats not alive

SECONDARY OUTCOMES:
Microvascular complications including renal anemia | Average time is 10 years
Macrovascular complications | Average time is 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Kyuzi Kamoi, MD, Principal Investigator — Nagaoka Red Cross Hospital
Locations (1):
- Nagaoka Red Cross Hospital, Nagaoka, Niigata, Japan

REFERENCES:
- [Result] Kamoi K, Miyakoshi M, Soda S, Kaneko S, Nakagawa O. Usefulness of home blood pressure measurement in the morning in type 2 diabetic patients. Diabetes Care. 2002 Dec;25(12):2218-23. doi: 10.2337/diacare.25.12.2218. PMID 12453964
- [Result] Kamoi K, Imamura Y, Miyakoshi M, Kobayashi C. Usefulness of home blood pressure measurement in the morning in type 1 diabetic patients. Diabetes Care. 2003 Aug;26(8):2473-5. doi: 10.2337/diacare.26.8.2473. No abstract available. PMID 12882886
- [Result] Kamoi K, Ito T, Miyakoshi M, Minagawa S. Usefulness of home blood pressure measurement in the morning in patients with type 2 diabetes: long-term results of a prospective longitudinal study. Clin Exp Hypertens. 2010 May;32(3):184-92. doi: 10.3109/10641960903254513. PMID 20504126